CLINICAL TRIAL: NCT01076829
Title: Inhibition of Absorption of Cytoxic Lipid Peroxidation Products and Abnormalities of Postprandial Endothelial Function by Spice Polyphenols Fed Together With High Fat Meat Patty in Men With Type 2 Diabetes Mellitus or Impaired Glucose Tolerance
Brief Title: Effects of a Spiced Meat Patty on Inflammation in Men With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, UCLA Center for Human Nutrition, Chief, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 08-11-023
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2013-12

CONDITIONS: Type II Diabetes Mellitus
Keywords: MDA; Spice
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spice patty (Active Comparator): hamburger meat cooked with spice mixture
  Interventions: Other: Spice polyphenols
- salt patty (Placebo Comparator): Subjects consume salt containing hamburger meat
  Interventions: Other: Spice polyphenols

INTERVENTIONS:
Other: Spice polyphenols — spice

SUMMARY:
Polyphenols belong to the largest group of secondary metabolites produced by plants, mainly, in response to biotic or abiotic stresses such as infections, wounding, UV irradiation, exposure to ozone, pollutants, and other hostile environmental conditions. It is thought that the molecular basis for the protective action of polyphenols in plants is their antioxidant and free radical scavenging properties. These numerous phenolic compounds are major biologically active components of spices, aromas, essential oils, and traditional medicines. In order to investigate the impact of spice polyphenols on postprandial flow-mediated dilation, nitric oxide, glucose, insulin, triglycerieds, oxidized LDL, and cytoxic lipid peroxidation products (MDA) levels in men with type 2 diabetes, the investigators propose to achieve the following specific aims using a randomized crossover study design:

1. To determine the effect of a ground beef patty meal with and without polyphenol-rich spices on postprandial levels of plasma oxidized LDL, triglycerides, insulin, glucose, and malondialdehyde (MDA).
2. To determine the effect of a ground beef patty meal with and without polyphenol-rich spices on postprandial levels of nitric oxide and flow-mediated dilation.
3. To determine the effect of a ground beef patty meal with and without a spice blend on MDA accumulation in urine.

This study will determine whether spice polyphenols exert a beneficial effect by inhibition of the absorption of lipotoxin MDA in males with type 2 diabetes mellitus.Men with diabetes mellitus type 2 have been selected for this study to enable assessment of markers of vascular health including nitric oxide in plasma and flow-mediated dilation. These findings may help to explain the potentially harmful effects of oxidizable fats found in foods and the important benefit of dietary polyphenols in ameliorating this potentially harmful effect.

DETAILED DESCRIPTION:
10 male subjects with type 2 diabetes mellitus who will be recruited based on inclusion and exclusion criteria. The study will be carried out in accordance with the guidelines of the Human Subjects Protection Committee of the University of California, Los Angeles. All subjects will give written informed consent before the study begins. After the screening visit, each subject will come to the Center for Human Nutrition on two 1-day test phases separated by at least one week. At each of phases, subjects will consume, in a random order, two different test meals consisting of either: a) a ground dark meat beef patty seasoned with salt only, or b) a ground dark meat beef patty seasoned with a spice mixture and salt. The subjects will be asked to avoid eating high fat meat meals and all spice products for 3 days before the day of each of the two experimental phases

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type II Diabetes Mellitus and currently being treated with oral medication but no insulin or glucose intolerant on no medications with a fasting blood sugar of > 110 mg/dl but less than 126 mg/dl fasting.
* Have an HbA1C lvel <9 % at Screening
* Male 35-70 years old
* Non-smokers, or smoke < 1 cigarette per day
* Must weigh a minimum of 110 pounds
* Willing to maintain normal activity and eating patterns for the duration of the study
* Willing to avoid meat, fish or poultry for three days on two occasions prior to the test procedure
* Consuming less than two alcoholic drinks per day
* Not taking dietary supplements
* No known allergy to beef, cloves, cinnamon, oregano, turmeric, cumin, rosemary, sage, red pepper, ginger, black pepper, paprika or garlic

Exclusion Criteria:

* Currently using insulin
* Abnormal liver function
* Currently taking steroidal drugs
* Known HIV positive or AIDS
* Chronic infectious disease
* Cancer treated within the past two years
* Participation in a therapeutic research study within 30 days of baseline
* Allergy to beef, cloves, cinnamon, oregano, rosemary, ginger, black pepper, paprika or tumeric
* History of hear failure with EF < 30, chronic renal failure with GFR < 30 ml/min
* Currently taking vasoactive medications such as but not limited to calcium channel blockers, nitrates, beta blockers, phosphodiesterase inhibitors
* History of Raynauds
* History of smoking within 5 years

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The protocol is designed to study the effect of spice on MDA production in hamburg meat | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- David Geffen School of Medicine, UCLA Center for Human Nutrtiion, Los Angeles, California, United States